CLINICAL TRIAL: NCT04971772
Title: SIGNATURE Study: Post-market, Randomized Controlled, Multicenter, Single Blinded Prospective Trial Investigating the Paclitaxel-Coated Balloon (Legflow DCB) Treatment Versus Uncoated Balloon Angioplasty Treatment for Femoro-popliteal Lesions.
Brief Title: SIGNATURE Study : DCB (Legflow) vs POBA in Fempop Arteries
Acronym: SIGNATURE
Status: Recruiting | Type: Observational
Sponsor: Cardionovum GmbH (Industry)
Collaborators: FCRE (Foundation for Cardiovascular Research and Education) (Other)
Responsible Party: Sponsor
Other Study IDs: FCRE-210621
Record Dates: First submitted 2021-07-20; First posted 2021-07-21 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Peripheral Arterial Disease; Superficial Femoral Artery Stenosis; Angiopathy, Peripheral
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DCB (Legflow .035") group: treatment with Drug Coated Balloon angioplasty with the Legflow .035" Paclitaxel Balloon Dilatation catheter.
- POBA group: treatment with standard POBA (uncoated) angioplasty (type and brand at the physician's discretion)

SUMMARY:
The aim of this study is to demonstrate the superiority in safety and efficacy of the Legflow DCB vs standard uncoated POBA in a randomized controlled (RCT) for treatment of patients with symptomatic peripheral artery disease (PAD) due to stenosis, restenosis or occlusion of the femoral and/or popliteal arteries.

ELIGIBILITY:
Inclusion criteria

* Patient is ≥18 years
* Patient has Rutherford Classification 2,3 or4.
* Patient has provided written informed consent and is willing to comply with study follow-up requirements.
* De novo stenotic or occlusive lesion(s) or non-stented restenotic or occlusive lesion(s) occurring >90 days after prior plain old balloon (POBA) angioplasty or >180 days after prior DCB treatment.
* Target lesion is located between the ostium of the SFA and the end of the P1 segment of the popliteal artery
* Target vessel diameter ≥ 4 mm and ≤ 7 mm
* Target lesion must be stenotic or occlusive lesion ≤ 150mm in length (one long lesion or tandem lesions) by investigator's visual estimate. [Note: tandem lesions must have a total length of ≤ 150 mm by visual estimate and be separated by ≤ 30 mm.]
* Target lesion must have angiographic evidence of ≥ 70 % stenosis by investigator's visual estimation
* Successful, uncomplicated crossing of the target lesion occurs when the tip of the guidewire is distal to the target lesion without the occurrence of flow-limiting dissection of perforation and is judged by visual inspection to be within the true lumen. Subintimal dissection techniques may be used if re-entry occurs above-the-knee (ATK) and without the use of re-entry devices.
* Target lesion is located at least 30mm from any stent if target vessel was previously stented.
* A patent inflow artery free from significant stenosis ((≥50% stenosis) as confirmed by angiography.
* At least one patent native outflow artery to the ankle or foot, free from significant stenosis (≥ 50 % stenosis) as confirmed by angiography.

Exclusion criteria:

* Acute Limb Ischemia
* Patient underwent an intervention involving the target vessel within the previous 90 days.
* Patient underwent any lower extremity percutaneous treatment in the ipsilateral limb using plain old balloon (POBA) angioplasty within the previous 90 days.
* Patient underwent a percutaneous transluminal angioplasty (PTA) of the target lesion using a DCB within the previous 180 days.
* Pregnant women or women who are intending to become pregnant.
* Patient has a life expectancy of less than 1 year
* Patient has a known allergy to contrast medium that cannot be adequately pre-medicated.
* Patient is allergic to all anti-platelet treatments
* Patient is receiving immunosuppressant therapy
* Patient has platelet count <100.000/mm3 or >700.000/mm
* Patient has history of gastrointestinal hemorrhage requiring a transfusion within 3 months prior to the study procedure
* Patient is diagnosed with coagulopathy that precludes treatment with systemic anticoagulation and/or dual antiplatelet therapy (DAPT)
* Patient has history of stroke within past 90 days
* Patient has history of myocardial infarction within the past 30 days.
* Patient is participating in an investigational drug or medical device study that has not completed primary endpoint(s) evaluation or that clinically interferes with the endpoints from this study.
* Patient has had any major (e.g. cardiac, peripheral, abdominal) surgical procedure or intervention unrelated to this study within 30 days prior to the index procedure or has planned major surgical procedure or intervention within 30 days of the index procedure
* An intervention in the contralateral limb, planned within 30 days post-index procedure
* Patient had previous bypass surgery of the target lesion
* Patient had previous treatment of the target vessel with thrombolysis or surgery
* Patient is unwilling or unable to comply with procedures specified in the protocol or has difficulty or inability to return for follow-up visits as specified by the protocol
* Target lesion involves an aneurysm or is adjacent to an aneurysm (within 5 mm)
* Target Lesion requires treatment with alternative therapy such as stenting, laser, atherectomy, cryoplasty, brachytherapy or re-entry devices
* Significant target vessel tortuosity or other parameters prohibiting access to the target lesion
* Presence of thrombus in the target vessel
* Iliac inflow disease requiring treatment, unless the iliac artery disease is successfully treated first during the index procedure. Success is defined as ≤ 30 % residual diameter stenosis without death or major complications.
* Presence of an aortic, iliac or femoral artificial graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral arterial disease in the SFA, eligible for treatment with the paclitaxel coated Legflow dilatation balloon catheter
Sampling Method: Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: | 12 months post-procedure
  The primary efficacy endpoint is time to clinically-driven target lesion revascularization (CD-TLR) at 12 months, defined as any reintervention at the target lesion due to symptoms OR drop of ankle brachial index (ABI) > 20 % OR ABI > 0.15 compared to the post-procedural ABI.
Device- and procedure-related death | 30 days post-procedure
  Primary Safety Endpoint:
  Freedom from device- and procedure-related death through 30 days post-index procedure;
Major target limb amputation and clinically-driven target vessel revascularization | 12 months post-procedure
  Primary Safety Endpoint:
  A composite of (2.1) time to major target limb amputation (above-the-ankle (ATA)) through 12 months post-procedure and (2.2) time to clinically-driven target vessel revascularization (CD-TVR) through 12 months post-index procedure

SECONDARY OUTCOMES:
Acute device success | during index procedure
  defined as successful delivery, balloon inflation, deflation and retrieval of the intact study device without burst below rated burst pressure
Acute procedural success | during index procedure
  Acute procedural success is defined as restoration of the target lesion with ≤30% residual stenosis in the final angiogram.
Secondary safety endpoint at discharge up to 30 days post-index procedure | 30 days post-operative
  Secondary safety endpoint is a composite of (3.1) freedom from all cause death (3.2) freedom from major target limb amputation (3.3) freedom from CD-TVR
Sustained clinical improvement at 6-, 12- and 24- months post-index procedure | 6, 12, 24-months post-procedure
  Clinical improvement is defined as a composite of (4.1) freedom from major target limb amputation, (4.2) freedom from TVR, (4.3) freedom from worsening target limb Rutherford class (compared to baseline) (4.4) freedom from decrease in target limb ankle brachial index (ABI) ≥0.15 (compared to baseline)
Major Adverse Events (MAEs) at 6-, 12- and 24-months post-index procedure | 6, 12, 24-months post-procedure
  MAEs are defined as composite of (5.1) all-cause death, (5.2) CD-TVR (5.3) major target limb amputation (5.4) thrombosis at the target lesion
Primary Patency at 6-, 12- and 24-months | 6, 12, 24-months post-procedure
  The primary patency is defined as a composite of (6.1) freedom from clinically-driven target lesion revascularization (CD-TLR)
  (6.2) freedom from binary restenosis (restenosis defined as duplex ultrasound (DUS) peak systolic velocity ratio (PSVR) ≥2.4 or ≥50% stenosis)
  • For discharge and 12-months: assessed by independent Core Lab
Target Lesion Revascularization at 6-, 12- and 24-months post-index procedure | 6, 12, 24-months post-procedure
  defined as a reintervention to maintain or restore the patency in the target lesion. TLR is clinically-driven (CD) when the TLR was needed due to symptoms or drop of ankle brachial index (ABI) of ≥20% or >0.15 when compared to post-procedure.
Target Vessel Revascularization at 6-, 12- and 24-months post-index procedure | 6, 12, 24-months post-procedure
  defined as a reintervention to maintain or restore the patency in the target vessel. TVR is clinically-driven (CD) when the TVR was needed due to symptoms or drop of ankle brachial index (ABI) of ≥20% or >0.15 when compared to post-procedure
Binary restenosis at 6-, 12- and 24-months | 6, 12, 24-months post-procedure
  defined as a restenosis confirmed by DUS PSVR ≥2.4 or ≥50% stenosis (For 12-month: assessed by Independent Core-Lab)
Major Target Limb Amputation at 6-, 12- and 24-months | 30- days, 6, 12, 24-months post-procedure
  defined as an amputation above the ankle (ATA) in the target limb
Thrombosis at the target lesion at 6-, 12- and 24-months | 6, 12, 24-months post-procedure
  Thrombosis at the target lesion at 6-, 12- and 24-months
All-cause death at 6-, 12- and 24-months | 30- days, 6, 12, 24-months post-procedure
  All-cause death at 6-, 12- and 24-months
Change in target limb Rutherford Classification from baseline to 6-, 12- and 24-months | 6, 12, 24-months post-procedure
  Change in Target Limb Rutherford Classification from baseline to 6-, 12- and 24-months
Change in Target Limb Resting ABI or TBI from baseline to 6-, 12- and 24-months | 6, 12, 24-months post-procedure
  Change in Target Limb Resting ABI or TBI from baseline to 6-, 12- and 24-months
Improvement of life quality according to the Walking Impairment Questionnaire (WIQ) and the EQ-5D Questionnaire to baseline at follow-up at 6-, 12- and 24-month. | 6, 12, 24-months post-procedure
  Improvement of life quality according to the Walking Impairment Questionnaire (WIQ) and the EQ-5D Questionnaire to baseline at follow-up at 6-, 12- and 24-month.
device- and procedure-related death | 30- days, 6, 12, 24-months post-procedure
  Freedom from device- and procedure-related death at discharge, 30 days, 6-, 12- and 24-months

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Sankt Gertrauden-Krankenhaus Berlin, Berlin
  - Medizinisches Versorgungszentrum Prof. Mathey, Prof. Schofer GmbH, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - SRH Klinikum Karlsbad-Langenseinbach GmbH, Karlsbad
  - St. Franziskus-Hospital GmbH, Münster
  - GRN-Klinik Weinheim, Weinheim

IPD SHARING:
Plan to Share IPD: No